CLINICAL TRIAL: NCT02227316
Title: A Prospective, Double Blind, Randomized, Placebo Controlled Study to Compare the Effectiveness of Intravenous Acetaminophen and Intravenous Ibuprofen in Reducing Post Procedural Pain in the Uterine Fibroid Embolization Procedure
Brief Title: Effectiveness of IV Acetaminophen and IV Ibuprofen in Reducing Post Procedural Pain in the UFE Procedure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Sponsor Name Pending (Industry)
Responsible Party: Principal Investigator, Cheryl Hoffman, MD., University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14000359
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Symptomatic Uterine Fibroids and Adenomyosis
Keywords: Uterine Fibroid Embolization; Pain; UFE; Fibroids; Adenomyosis; Bleeding; IV Acetaminophen; IV Ibuprofen; Menorrhagia; Leiomyoma; Patient Satisfaction
MeSH Terms: conditions — Adenomyosis; Pain; Leiomyoma; Hemorrhage; Menorrhagia; Patient Satisfaction | interventions — Ibuprofen; Uterine Artery Embolization; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intravenous Ibuprofen (Experimental): Ibuprofen 800mg IV piggyback and Saline IVP q 6 hours x 4 during uterine fibroid embolization
  Interventions: Drug: IV Ibuprofen
- Intravenous acetaminophen (Experimental): Acetaminophen 1 gram IV piggyback and Saline IVP q6 hours x 4 during uterine fibroid embolization
  Interventions: Drug: IV Acetaminophen
- IV ibuprofen/IV acetaminophen (Experimental): Ibuprofen 800 mg/ Acetaminophen 1 gram IV piggyback and Saline IVP 6 hours x 4 during uterine fibroid embolization
  Interventions: Drug: IV Ibuprofen; Drug: IV Acetaminophen
- Intravenous placebo/Intravenous placebo (Active Comparator): Saline/Saline IV piggyback and IVP Ketorolac 30 mg q6 hours x 4 during uterine fibroid embolization
  Interventions: Drug: Intravenous placebo/Intravenous placebo

INTERVENTIONS:
Drug: IV Ibuprofen — Uterine fibroid embolization
  Other Names: Uterine artery embolization
  Arms: IV ibuprofen/IV acetaminophen; Intravenous Ibuprofen
Drug: IV Acetaminophen — Uterine fibroid embolization
  Other Names: Uterine artery embolization
  Arms: IV ibuprofen/IV acetaminophen; Intravenous acetaminophen
Drug: Intravenous placebo/Intravenous placebo — Uterine fibroid embolization
  Other Names: Uterine artery embolization
  Arms: Intravenous placebo/Intravenous placebo

SUMMARY:
The uterine fibroid embolization (UFE) procedure is a treatment option for abnormal heavy menstrual bleeding and/or bulk symptoms associated with uterine fibroids and adenomyosis. Post UFE procedural pain and nausea are expected events. These symptoms are treated with current standard of care medications, including opiates.

Intra procedure pain medications include midazolam, fentanyl and hydromorphone. Some centers include nonsteroidal anti-inflammatory medications (NSAIDS), including oral ibuprofen and IV ketorolac. Post procedural pain control is centered on a hydromorphone patient-controlled analgesia (PCA) infusion pump, as well as a NSAID regimen. Intra procedure and post procedure nausea control medications include a transcutaneous scopolamine patch and IV anti-nausea medications such as ondansetron and prochlorperazine.

This study is being conducted to compare two new medications for pain, IV ibuprofen and IV acetaminophen, administered for 24 hours following UFE. The primary safety objective of non-inferiority will be met and the primary efficacy objective of superiority, decreased pain and nausea, will be accessed when compared to current standard of care regimens.

This is a 4 arm, double blind, randomized, controlled study. All patients will receive standard of care baseline pain medications, including IV midazolam, fentanyl and hydromorphone intra procedure, followed by a hydromorphone PCA infusion pump post procedure. The 4 arms will include: [ Arm 1] IV ibuprofen/IV placebo, [Arm 2] IV acetaminophen/IV placebo, [Arm 3] IV ibuprofen/IV acetaminophen, and [arm 4] IV placebo/IV placebo. These medications will be given during the procedure and extended over a 24 hour stay.

Arm 4 (IV placebo/IV placebo) would replicate current standard of care, and therefore will include IV push (IVP) ketorolac, which would be given at the end of the procedure and be continued every 6 hours for the 24 hour stay. An IVP of saline will be given as a control every 6 hours for the 24 hour stay to arms 1, 2 and 3. Pain and nausea will be measured at intervals prior to the procedure, throughout the stay and at 2 weeks post procedure.

DETAILED DESCRIPTION:
A prospective, double blind, randomized controlled trial evaluating the effects of two new IV medications, IV ibuprofen and IV acetaminophen, on standard of care pain and anti-emetic management in Uterine Fibroid Embolization patients.

1. Four arm, double blind, randomized controlled study: all patients will receive standard of care baseline pain medications, including IV midazolam, fentanyl and hydromorphone during the procedure, followed by a hydromorphone PCA infusion pump during their recovery. The four arms will include an IV ibuprofen/IV placebo, an IV acetaminophen/IV placebo, an IV ibuprofen/IV acetaminophen, and a control arm (IV placebo/IV placebo). The same amount of normal saline will be substituted for the experimental treatments if the patient receives the placebo. These medications will be given during the procedure and extended over a 24 hour recovery period. The medications given will be blinded to the patient, the administrator, and the surveyor.
2. The placebo/placebo arm would replicate current standard of care, and therefore include IV push (IVP) ketorolac, which would be given at the end of the procedure and be continued for 24 hours at q6hour dosing. An IVP of saline would be given as a control for 24 hours at q6hour dosing to the other three arms.
3. Dosage of medications will be standardized based on formulary indications: IV Ketorolac 30 mg/dose IVP, acetaminophen 1 gram/dose IV piggy back over 15 minutes every 6 hours, ibuprofen 800 mg/dose IV piggy back over 30 minutes every 6 hours.
4. Variables measured: mean and maximum pain (VAS score at 0 hours, 6 hours, discharge and 2 weeks post procedure), opioid requirements, mean and maximum nausea (VAS score at 0 hours, 6 hours, discharge and 2 weeks post procedure), anti-emetic medication requirements.

   Weighted sum of pain intensity differences, with pain intensity measured on VAS over 24 hours (SPID24) will be used as a primary outcome. Satisfaction scores will be measured at 24 hours using the validated APS-POQ-R questionnaire (6).
5. Other variables recorded: Age, height, weight, history of postoperative nausea and vomiting or motion sickness, diagnosis, uterine volume, dominant fibroid size, arteries embolized, presence of prominent ovarian arteries, volume of particle used, fluoroscopy time for the procedure.
6. Technical parameters, which would remain constant, include: pre procedure and 6 month follow up MRI contrast with gadolinium which is standard of care, embolization using 500-700 micron Embospheres (with limited use of 700-900 micron Embospheres), IV hydration with 0.9% normal saline, antibiotics (IV ciprofloxacin 400 mg every 12 hours, IV metronidazole 500 mg every six hours), urinary catheter placement, lower extremity compression devices, and early ambulation.
7. In the interim analysis, the investigators will have 40 subjects in total with unequal randomization ratio of 1:1:4:4. Additional subjects will be enrolled for a total of 35 subjects per arm for the final analysis (sum total N=140)

ELIGIBILITY:
Inclusion Criteria:

1. Patients being considered for UFE including bleeding and/or bulk symptoms.
2. Women of all ethnicities
3. Ages 21-60

Exclusion Criteria:

1. Patients with current malignancy receiving treatment
2. Women who are pregnant
3. Cognitive impairment
4. Clinically significant kidney disease
5. Clinically significant liver disease
6. Any recent history of gastrointestinal bleed or ulcer
7. Weight less than 50 kg (medication dosing requirements change below 50 kg)
8. Women with a body mass index (BMI) equal to or over 50 (with other co-morbidities)
9. Known allergy or hypersensitivity to NSAID or acetaminophen
10. Administration of acetaminophen, NSAID, narcotic or any other analgesic less than 6 hours prior to UFE procedure
11. Any chronic use of pain medications including acetaminophen, NSAID, narcotic or analgesic
12. Patients who cannot or choose not to consent to participate in the study

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl H Hoffman, MD, Principal Investigator — University of California, Los Angeles; Jonathan S Jahr, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Santa Monica/UCLA Medical Center and Orthopaedic Hospital, Santa Monica, California

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were excluded before assignment to groups.
Groups:
- Intravenous Ibuprofen: Ibuprofen 800mg IV piggyback and Saline IVP q 6 hours x 4.
  IV Ibuprofen
- Intravenous Acetaminophen: Acetaminophen 1 gram IV piggyback and Saline IVP q6 hours x 4
  IV Acetaminophen
- IV Ibuprofen/IV Acetaminophen: Ibuprofen 800 mg/ Acetaminophen 1 gram IV piggyback and Saline IVP 6 hours x 4
  IV Ibuprofen
  IV Acetaminophen
- Intravenous Placebo/Intravenous Placebo: Saline/Saline IV piggyback and IVP Ketorolac 30 mg q6 hours x 4
  IV Placebo
Period: Overall Study
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Started | 4 | 4 | 16 | 16
Completed | 4 | 4 | 16 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo | Total
Number analyzed (Participants) | 4 | 4 | 16 | 16 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 16 | 16 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.96 (3.22) | 45.24 (6.31) | 44.33 (4.32) | 44.49 (4.12) | 44.25 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 16 | 16 | 40
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 16 | 16 | 40

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Maximum Pain Intensity Change Over 24 Hours With the Addition of IV Acetaminophen and IV Ibuprofen
Description: Primary efficacy objective is to compare the change in maximum level of pain experienced by patient over 24 hours between IV acetaminophen and IV ibuprofen (alone and in combination), and the current standard of care medication regimen. This comparison will be measured using a visual analog scale (VAS) from 0 to 10, 0 signifying no pain and 10 signifying the worst possible pain. The scores reported are the mean of all patients' VAS scores in each respective category.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Number analyzed (Participants) | 4 | 4 | 16 | 16
units on a scale | 6.48 (0.21) | 7.27 (1.17) | 6.16 (0.59) | 5.30 (1.45)

2. Primary Outcome: Evaluation of Mean Pain Intensity Over 24 Hours With the Addition of IV Acetaminophen and IV Ibuprofen
Description: Primary efficacy objective is to compare the change in mean pain intensity score over 24 hours between IV acetaminophen and IV ibuprofen (alone and in combination), and the current standard of care medication regimen. This comparison will be measured using a visual analog scale (VAS) from 0 to 10, 0 signifying no pain and 10 signifying the worst possible pain. The scores reported are the mean of all patients' VAS scores in each respective category.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Number analyzed (Participants) | 4 | 4 | 16 | 16
units on a scale | 4.52 (1.19) | 4.22 (0.92) | 3.90 (1.39) | 3.34 (1.07)

3. Secondary Outcome: Mean Nausea Intensity
Description: Assessment of mean nausea by mean of VAS scores over a 24-hour period. VAS score is measured using a scale of 0 to 10, 0 signifying no nausea and 10 signifying the worst possible nausea. The scores reported are the mean of all patients' VAS scores in each respective category.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Number analyzed (Participants) | 4 | 4 | 16 | 16
units on a scale | 1.52 (0.91) | 3.20 (0.80) | 3.59 (0.35) | 2.38 (0.79)

4. Secondary Outcome: Opioid Consumption
Description: Mean opioid consumption in morphine equivalents over 24 hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Morphine equivalent
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Number analyzed (Participants) | 4 | 4 | 16 | 16
Morphine equivalent | 75.75 (38.53) | 69.63 (7.30) | 48.44 (22.42) | 62.28 (35.02)

5. Secondary Outcome: Anti-Emetic Consumption
Description: Mean dose of anti-emetic medication in milligrams given over 24 hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Milligrams
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Number analyzed (Participants) | 4 | 4 | 16 | 16
Milligrams | 16.00 (8.64) | 19.50 (7.30) | 22.25 (7.72) | 19.50 (11.76)

6. Secondary Outcome: Maximum Nausea Intensity
Description: Assessment of maximum level of nausea experienced by patient, by mean of VAS scores over a 24-hour period. VAS score is measured using a scale of 0 to 10, 0 signifying no nausea and 10 signifying the worst possible nausea. The scores reported are the mean of all patients' VAS scores in each respective category.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Number analyzed (Participants) | 4 | 4 | 16 | 16
units on a scale | 5.62 (2.88) | 5.25 (1.07) | 6.41 (0.94) | 3.71 (0.29)

ADVERSE EVENTS:
Arm/Group | Intravenous Ibuprofen | Intravenous Acetaminophen | IV Ibuprofen/IV Acetaminophen | Intravenous Placebo/Intravenous Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes